CLINICAL TRIAL: NCT01762085
Title: A Prospective Study of Recurrence Risk in Diabetic Foot Ulceration After Nerve Decompression
Brief Title: Nerve Decompression for Ulcer Recurrence Avoidance (DURA)
Acronym: DURA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association of Extremity Nerve Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WIRB 20122035; Nerve DURA (Other Grant/Funding Number: AENS/ENRF)
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Diabetic Ulcer of Plantar Aspect of Left Foot; Diabetic Ulcer of Plantar Aspect of Right Foot; Diabetic Polyneuropathy
Keywords: neuropathic diabetic foot ulcer; nerve decompression surgery
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Decompression, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healed DFU control arm (Placebo Comparator): clinic-specific usual "best care"
- healed DFU surgical intervention (Experimental): clinic-specific "best care" plus nerve decompression at 4 known sites of lower leg fibro-osseous entrapment
  Interventions: Procedure: nerve decompression

INTERVENTIONS:
Procedure: nerve decompression — surgical decompression involves surgical division or incision of perineural fibrous or fibro-osseous tunnel tissues which pinch, choke, compress or sharply deviate nerve trunks.
  Other Names: nerve release; external neurolysis; surgical decompression
  Arms: healed DFU surgical intervention

SUMMARY:
Anecdotal reports and scientific literature suggest that the risk of recurrence of diabetic foot ulcers can be minimized by nerve decompression procedures at anatomic sites of nerve pinching and entrapment. Historical risk of 25% annually has been reported to decrease by >80% to under 5% yearly. Since an open wound precedes the large majority (85%) of amputations in diabetes, avoidance of ulcer recurrences is important. This study tests the current academic opinion that nerve decompression will not decrease ulcer recurrence risk. Null hypothesis: nerve decompression will not decrease diabetic foot ulcer recurrence risk.

DETAILED DESCRIPTION:
Diabetes patients with a recently healed, non-ischemic plantar diabetic foot ulcer will be randomized to "best care" standard post-ulcer treatment or to best care plus bilateral nerve decompression by external neurolysis at 4 fibro-osseous tunnel sites in the leg and foot. Comparison of the control group with standard care to the surgical intervention group will be made for subsequent appearance of a plantar foot ulcer and ulcer recurrence risks will be calculated. Additional subjective and objective secondary outcomes will be monitored. Null hypothesis: nerve decompression will not decrease diabetic foot ulcer recurrence risk.

If protection against ulcer occurrence were to be confirmed, a change in the treatment paradigm for diabetic neuropathy and foot ulcer could be appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 Diabetes Mellitus
* Diabetic sensorimotor peripheral neuropathy
* Recently healed plantar neuropathic Diabetic Foot Ulcer (< 18 months)
* At least one palpable foot or ankle pulse or ABI>0.8 bilaterally.
* Recent Hgb A1c < 9.0%
* Ankle edema absent or mild

Exclusion Criteria:

* Ischemic peripheral vascular disease or ankle-brachial index (ABI)<0.8
* History of peripheral vascular arterial surgery
* History of peripheral nerve or lumbar disc surgery
* alcohol abuse(more than 2 drinks/day)
* untreated thyroid disorders
* B12 or Folate deficiency
* spondyloarthropathies
* hepatic disease
* advanced renal disease
* current lumbosacral radiculopathy or nerve compression
* toxin exposure including chemotherapeutic agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
occurrence of plantar foot ulceration wound | 2 years post-enrollment or post-op
  Non- traumatic pressure wound or ulcer appearance during the study.

SECONDARY OUTCOMES:
occurrence of delayed wound healing | 3 months post nerve decompression
  failure of surgical wound to heal primarily, without local infection signs of swelling, heat, redness, and pain
Visual Analog Pain Score | 2 years
  Patient report of pain level

OTHER OUTCOMES:
any amputation | 24 months, 2 years
  surgical removal of any part of the lower extremity, including toe
surgical wound infection | 3 months
  swelling, redness, or heat, with pain after surgery
non-surgical foot infection | 24 months
  foot swelling, redness, pain, and heat not subsequent to operation; or occurring in an operated leg >90 days post-op
measures of diabetic peripheral neuropathy (DPN) | 2 years
  Michigan Neuropathy Symptom Index; Pain visual analog pain scale (VAPS); sensibility to vibration, light touch, 2-point discrimination; deep tendon reflex
analgesic usage | 2 years
  patients will log use of analgesic medications and changes in use.
SPY Indocyanine green circulation evaluation | pre-opo, post-op, study end
  This intravenous injection and non-invasive scan evaluation may indicate whether relief of nerve entrapment will alter macro or microcirculation
Incidence of falls during the study | 2 years
  Prior history of falls will be defined and changes in risk of new falls in control and intervention groups. Balance has been reported to improve after nerve decompression.

CONTACTS AND LOCATIONS:
Overall Officials: D. Scott Nickerson, MD, Study Director — NE Wyoming Wound Care Center, consultant; Stephen L. Barrett, DPM, Principal Investigator — Barrett Foot & Ankle Institute
Locations (6):
- United States (6):
  - Barrett Foot & Ankle Institute, Phoenix, Arizona
  - Richard P. Jacoby, Scottsdale, Arizona
  - Southern Arizona Limb Salvage Alliance,, Tucson, Arizona
  - Andrew Rader, DPM, Jasper, Indiana
  - Damien Dauphinee, Denton, Texas
  - Maria Buitrago, DPM, Houston, Texas

REFERENCES:
- [Background] Aszmann O, Tassler PL, Dellon AL. Changing the natural history of diabetic neuropathy: incidence of ulcer/amputation in the contralateral limb of patients with a unilateral nerve decompression procedure. Ann Plast Surg. 2004 Dec;53(6):517-22. doi: 10.1097/01.sap.0000143605.60384.4e. PMID 15602245
- [Background] Dellon AL. Preventing foot ulceration and amputation by decompressing peripheral nerves in patients with diabetic neuropathy. Ostomy Wound Manage. 2002 Sep;48(9):36-45. PMID 12271732
- [Background] Dellon AL. Neurosurgical prevention of ulceration and amputation by decompression of lower extremity peripheral nerves in diabetic neuropathy: update 2006. Acta Neurochir Suppl. 2007;100:149-51. doi: 10.1007/978-3-211-72958-8_32. PMID 17985566
- [Background] Nickerson DS. Low recurrence rate of diabetic foot ulcer after nerve decompression. J Am Podiatr Med Assoc. 2010 Mar-Apr;100(2):111-5. doi: 10.7547/1000111. PMID 20237362
- [Background] Dellon AL, Muse VL, Nickerson DS, Akre T, Anderson SR, Barrett SL, Biddinger KR, Bregman PJ, Bullard BP, Dauphinee DM, DeJesus JM, DeJesus RA, Ducic I, Dunkerly J, Galina MR, Hung V, Ichtertz DR, Kutka MF, Jacoby RP, Johnson JB, Mader DW, Maloney CT Jr, Mancuso PJ, Martin RC, Martin RF, McDowel BA, Rizzo VJ, Rose M, Rosson GD, Shafiroff BB, Steck JK, Stolarski RG, Swier P, Wellens-Bruschayt TA, Wilke B, Williams EH, Wood MA, Wood WA, Younes MP, Yuksel F. Prevention of ulceration, amputation, and reduction of hospitalization: outcomes of a prospective multicenter trial of tibial neurolysis in patients with diabetic neuropathy. J Reconstr Microsurg. 2012 May;28(4):241-6. doi: 10.1055/s-0032-1306372. Epub 2012 Mar 12. PMID 22411624
- [Background] Dellon AL. A cause for optimism in diabetic neuropathy. Ann Plast Surg. 1988 Feb;20(2):103-5. doi: 10.1097/00000637-198802000-00001. No abstract available. PMID 3355053
- [Background] Dellon AL. Treatment of symptomatic diabetic neuropathy by surgical decompression of multiple peripheral nerves. Plast Reconstr Surg. 1992 Apr;89(4):689-97; discussion 698-9. PMID 1546082
- [Background] Rankin TM, Miller JD, Gruessner AC, Nickerson DS. Illustration of Cost Saving Implications of Lower Extremity Nerve Decompression to Prevent Recurrence of Diabetic Foot Ulceration. J Diabetes Sci Technol. 2015 Jul;9(4):873-80. doi: 10.1177/1932296815584796. Epub 2015 Jun 8. PMID 26055081